CLINICAL TRIAL: NCT06134921
Title: The Effects of Bilateral-Transcranial Electrical Stimulation (tES) on Cortical Activity, Motor Performances, and Cognitive Function in Sub-Acute and Chronic Stroke Individuals
Brief Title: Effects of Transcranial Electrical Stimulation in Stroke Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU-CIRB 2023/288.1509
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke; Chronic Stroke; Subacute Stroke
Keywords: transcranial electrical stimulation; stroke; electroencephalography; rehabilitation
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS and conventional physical therapy program (Experimental): Participants will receive Active tDCS for 30 minutes prior conventional physical therapy program. They will be asked to perform this combination therapy for 15 sessions, occurring three times a week for five weeks.
  Interventions: Device: transcranial direct current stimulation (Active); Other: Conventional physical therapy program
- Active tACS and conventional physical therapy program (Experimental): Participants will receive Active tACS for 30 minutes prior conventional physical therapy program. They will be asked to perform this combination therapy for 15 sessions, occurring three times a week for five weeks.
  Interventions: Device: transcranial alternating current stimulation (active); Other: Conventional physical therapy program
- Sham stimulation and conventional physical therapy program (Sham Comparator): Participants will receive sham stimulation for 30 minutes prior conventional physical therapy program. They will be asked to perform this combination therapy for 15 sessions, occurring three times a week for five weeks.
  Interventions: Device: transcranial electrical stimulation (sham); Other: Conventional physical therapy program

INTERVENTIONS:
Device: transcranial direct current stimulation (Active) — Electrode placement based on the international 10 - 20 electroencephalography electrode system for the cathodal electrode will be applied over the contralesional hemisphere. In contrast, an anodal electrode will be applied over the ipsilesional hemisphere on the primary motor cortex (C3 or C4). Participants will be asked to sit comfortably during stimulation.
  In the Active-tDCS group, participants will receive real tDCS with intensity 2.0 mA for 30 minutes, with a 30-second ramp-up and ramp-down.
  Other Names: tDCS (Active); innk; Neurophet, Korea
  Arms: Active tDCS and conventional physical therapy program
Device: transcranial alternating current stimulation (active) — Electrode placement based on the international 10 - 20 electroencephalography electrode system for the cathodal electrode will be applied over the contralesional hemisphere. In contrast, an anodal electrode will be applied over the ipsilesional hemisphere on the primary motor cortex (C3 or C4). Participants will be asked to sit comfortably during stimulation.
  Other Names: tACS (Active); innk; Neurophet, Korea
  Arms: Active tACS and conventional physical therapy program
Device: transcranial electrical stimulation (sham) — Electrode placement based on the international 10 - 20 electroencephalography electrode system for applied the cathodal electrode will be applied over the contralesional hemisphere. In contrast, an anodal electrode will be applied over the ipsilesional hemisphere on the primary motor cortex (C3 or C4). Participants will be asked to sit comfortably during stimulation.
  In the Sham group, participants will receive sham stimulation with intensity 2.0 mA for 1 minute, with a 30-second ramp-up and ramp-down, and no stimulation until the end of 30 minutes of stimulation. Electrodes will remain for 30 minutes.
  Other Names: Sham stimulation; innk; Neurophet, Korea
  Arms: Sham stimulation and conventional physical therapy program
Other: Conventional physical therapy program — A conventional physical therapy program will be provided after 30 minutes of stimulation immediately. The program will be provided for both upper and lower limbs which consist of stretching exercise, active exercise, and functional exercise.

SUMMARY:
The present study will use transcranial electrical stimulation (tES) with conventional physical therapy in sub-acute (at least 2 weeks after stroke onset) to chronic stroke within 2 years to investigate the effect on cortical activity and upper and lower limb motor function. The findings may support the usage of tES for improving brain activity and motor function in a clinic setting.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and disability in the world. The prevalence of stroke is high in developing countries; for example in Thailand, stroke is one of a leading cause of death and disability. The estimate prevalence among adults aged 45 years and older is 1.88%, and the mortal rate of stroke is still has continued to increase over the past 5 years. Globally, 87 percent of stroke people have suffered from ischemic stroke while 13% suffered from hemorrhagic stroke. Fifty-seven percent stroke cases remains disability reported by the world stroke organization. Motor impairment is a major limit post-stroke and it affects activities in daily life. Cognitive impairments (i.e., executive function, attention, and memory) are commonly observed in post-stroke survivors which may lead decrease in functional capacity and affects the efficacy of rehabilitation in stroke.

Stroke is defined as a sudden neurological explosion caused by impaired perfusion through the blood vessels to the brain. Ischemic stroke is caused by deficient blood flow and oxygen supply to the brain, while, hemorrhagic stroke is caused by bleeding or leaky blood vessels, resulting in cell death. After-stroke, cortical excitability decreases in the ipsilesional hemisphere and increases in the contralesional hemisphere. Consequently, there is an imbalance in the interhemispheric inhibition (IHI) between both hemispheres. The onset of IHI imbalance in stroke patients remains unclear, although the occurrence of motor impairment since the onset. However, the IHI imbalance is remained throughout stroke life. The imbalance of IHI was found to be negatively correlated with stroke motor recovery; a greater imbalance was associated with a poorer motor performance. IHI imbalance is not a cause of poor motor recovery, but instead might be the consequence of underlying recovery processes.

An electroencephalography (EEG) is the non-invasive measurement tool with high temporal resolution, which can detect a summary of the postsynaptic electrical signals of pyramidal neurons in the cortical layers. EEG is a useful measurement after stroke. Several metrics have been found to be related to recovery across all stroke phases. A recent review in 2022 reported that brain symmetry index (BSI) and spectral power are the most efficacious metrics to use to predict stroke recovery. BSI is one of the more popular EEG-derived parameters use to quantify the mean spectral asymmetry between the two hemispheres. It has a normal range of 0 to 1, where 0 indicates perfect symmetry, while 1 indicates maximal asymmetry. BSI was significantly higher in stroke patients indicating brain asymmetry compared with healthy controls Van Putten and Tavy demonstrated in acute ischemic stroke people that BSI was unchanged within 24 hours post-stroke, however it had a positive correlation between the National Institutes of Health Stroke Scale (NIHSS); a higher impairment, a higher brain asymmetry. It was reported that higher BSI value in the acute to sub-acute phase were associated with lower motor performance in 4 weeks later implying that BSI could possibly aid in prognostication of motor outcome during stroke recovery phase. Moreover, spectral power analysis in stroke individuals showed fluctuation of brain oscillation caused by cell death such as an increase of low frequency power (delta and theta) in the ipsilesional hemisphere that occurred as early as one minute after stroke, whereas high frequency power (alpha and beta) were decreased. An increase in delta activity post-stroke was also negatively corelated to cognitive functioning. Cortical activity in recovery phase can represent motor recovery and cognitive function post-stroke. An increase of high-frequency brain wave (i.e. beta band) is related to improve motor recovery in subacute and chronic phases of stroke. In addition, increase of alpha band and decrease of delta band correlated with improve cognitive function in stroke survivors.

Motor recovery post-stroke rapidly increase within first 3 months (acute to early subacute phase) and less significant recovery subsequently in late-subacute (3-6 months), then, spontaneous recovery is leading to a stable at its limit in chronic phase (>6 months), but the recovery can expand up to 2 years post-stroke after receiving rehabilitation. Therefore, the rehabilitation can enhance stroke recovery beyond spontaneous recovery in the subacute and chronic phases. There are 2 factors influencing stroke recovery: 1) intrinsic factors which are age, sex, stroke onset, stroke type, severity, co-morbidities, socioeconomic status, and genetic profiles, 2) extrinsic factors such as caregiver support, pharmacology, and rehabilitation program in which consists of bottom-up and top-down approaches. Rehabilitation post-stroke is recommended to enhance recovery and reduce long-term disability. The guideline of American Stroke Association (ASA) has recommended that patients with stroke required therapeutic intervention of at least 3 times per week for 20-60 min per session.

Non-invasive brain stimulation (NIBS) i.e., transcranial Electrical stimulation (tES) is a top-down approach that has been recommended to use as an add-on intervention in rehabilitation post-stroke. The most common tES techniques used in research are 1) transcranial Direct Current Stimulation (tDCS) and 2) transcranial Alternating Current Stimulation (tACS). The difference between these two tES techniques is the current forms elicited.

1. tDCS delivers weak direct current to modulate cortical excitability with polarity-specific effects. Within dose limited, anodal tDCS enhances cortical excitability while cathodal tDCS decreases it. There are several studies reported the effect of tDCS on physical and cognitive performance in healthy subjects as well as in people with neurological disorders. To promote rebalancing of IHI, tDCS is used by applying anodal electrode over the ipsilesional hemisphere and cathodal electrode over the contralesional hemisphere simultaneously, called dual- or bilateral-tDCS. Many meta-analysis and individuals studies demonstrated that bilateral-tDCS over the primary motor cortex (M1) was more efficient for improving upper and lower limbs motor performances compared to other montages. Most of previous studies employed different intensities of 2 mA with duration of stimulation for 20 minutes. However, a recent meta-analysis suggested that a stimulation duration greater than 20 minutes to increase stimulation duration and number of stimulation session during 15 - 20 sessions were effective to enhance the effect of tDCS on motor function. For cognitive function, a recent meta-analysis reported the positive effect of tDCS applied over the dorsolateral prefrontal cortex (DLPFC) on cognitive function recovery compared with sham in stroke population. A previous study reported that tDCS targeting M1 combined with motor training could improve motor and cognitive performance, although the effect may less compared with targeting DLPFC.
2. tACS delivers alternating electrical current to modulate cortical excitability and endogenous brain oscillation with the frequency-specific. The activity of alpha (8-12 Hz) and beta (13-30 Hz) frequency is prominent in the human sensorimotor cortex during the resting-state. From a meta-analysis, tACS delivered at the beta frequency range could increase cortical excitability of the primary motor cortex. This effect is particularly pronounced when stimulation intensity was above 1 mA. In healthy populations, some studies have shown that a beta-tACS applied over the M1 could improve motor learning, and a greater effect was found when compared to alpha-tACS. Same observation was reported in stroke population, beta-tACS (20 Hz) at 1 mA induced greater modulation effects compared to alpha-tACS (10 Hz at 1 mA in the motor-related regions. Ten-session of tACS at 2mA over the M1 of the affected hemisphere with gait training could improve gait performance in individuals with chronic stroke. tACS appears to have potential for motor recovery post-stroke as other NIBS, but relevant numbers of randomized controlled trials (RCT) in stroke population are very limited compared to those of tDCS. Both tDCS and tACS are portable, easy to operate and induce only mild adverse effects. To now, there are few studies comparing the effects of tDCS with tACS. In terms of efficacy in cortical excitability alteration, with similar stimulation patterns (1.0 mA and 10 min), tACS significantly increased cortical excitability compared with sham in healthy subjects, however tDCS was not greater over sham. In term of motor performance, both beta-tACS (20 Hz) and anodal-tDCS over the M1 could increase reaction time in healthy subjects, with no significant difference on retrieval. However, in people with mild cognitive impairment, it was shown that tACS (40 Hz) applied over the DLPFC at 2 mA increase beta activity and cognitive function in comparison with 2 mA-tDCS and sham. tACS appeared to be superior to tDCS in improving cognitive outcomes.

Up to now, there is no study comparing the effects of tDCS and tACS in stroke population, especially on motor performance. To improve motor performance, the M1 is the most common target of electrical stimulation. Moreover, M1 stimulation together with motor training has been reported to improve motor and cognitive performance, The present study will investigate the effects of tDCS and tACS applied over the M1 combined with physical therapy on cortical activity, motor and cognitive outcomes in individuals with stroke in sub-acute and chronic phase within 2 years post stroke. Both tES techniques will be combined with conventional physical therapy for 15 sessions (3 days per week, 5 weeks) following by motor training as recommended by ASA. Cortical activity will be assessed by EEG and served as a primary outcome. Absolute spectral power of each frequency bands (alpha, beta, delta, theta) will be analyzed. Moreover, analysis of brain activity will be focused on brain symmetry index (BSI) which represents the balance between the contralesional and the ipsilesional hemispheres. Clinical outcomes will be served as a secondary outcome, for upper limb performance evaluations will consist of Fugl-Meyer assessment of upper (FMA-UE) and Wolf Motor Function Test (WMFT). For lower limb performance will be Fugl-Meyer assessment of lower (FMA-LE) and Timed Up and Go test (TUG). Five Time Sit to Stand (FTST), gait analysis and balance by using Zebris Force Distribution Measurement-T software and platform (FDM). Cognitive function will be examined by Montreal Cognitive Assessment (MoCA) in Thai version. All outcomes will be assessed at before-, post-intervention and 1-month and 3-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke individuals aged 18 - 80 years.
2. A first-ever unilateral ischemic or hemorrhagic stroke.
3. Stroke onset from at least 2 weeks - 2 years.
4. Having modified Rankin scale (mRS) 1-4
5. Ability to communicate, follow, and understand the instruction.

Exclusion Criteria:

1. Presence of any neurological antecedent, unstable medical conditions or condition that may increase risk of stimulation such as epilepsy and seizure, and history of brain surgery.
2. Presence of metal implantation, intracranial shunt, cochlear implantation, or cardiac pacemakers.
3. Presence of opened wound or infectious wound around the scalp.
4. Moderate pain in any joint of the upper or lower paretic limb (numerical pain rating score > 4/10).
5. History of receiving non-invasive brain stimulation within the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Absolute power | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  The raw data from electroencephalography (EEG) in 5-min of eye-opened and eye-closed conditions converted to the power distribution of brain waves in different frequencies (i.e., delta, theta, alpha, and beta) by using Fast Fourier Transformation (FFT)
Brain symmetry index (BSI) | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  The data from the absolute power will be used to calculate brain symmetry value ranged from 0-1( 0 represents perfect symmetry and 1 represents maximal asymmetry).

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) of upper and lower extremities | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  The FMA is used to quantify motor impairment and recovery post-stroke. The participants will use their unaffected side to perform first, and then subsequently perform their affected side in each movement 3 times. The best movement will be scored.
Timed Up and Go test | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Participants wear regular footwear and if they have normally used gait aid, it is allowed to use in the test. The test measures the time taken when the participants stand up from the chair, walk at normal pace for 3 meters, turn around, walk back for 3 meters, and then sit on a chair.
Five-Time Sit to Stand Test | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  The participants sit with the back lean against the chair, stand up and sit down 5 times as quickly as possible while keeping arm crossed throughout the test.
Spatiotemporal gait variables | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze the gait cycle. The force plate detects the force and weight bearing of the patient's feet and then calculates as step length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Spatiotemporal gait variables | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze the gait cycle. The force plate detects the force and weight bearing of the patient's feet and then calculates as stride length in centimeters (cm).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Spatiotemporal gait variables | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze the gait cycle. The force plate detects the force and weight bearing of the patient's feet and then calculates as single limb support (%).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Spatiotemporal gait variables | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze the gait cycle. The force plate detects the force and weight bearing of the patient's feet and then calculates as cadence (steps/min)
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Spatiotemporal gait variables | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  Force distribution measurement (FDM; The WinFDM and platform, Zebris Medical GmbH, Germany) will be used to analyze the gait cycle. The force plate detects the force and weight bearing of the patient's feet and then calculates as gait velocity (m/s).
  Participants will walk 3 meters per trial on a platform and be assessed 5 times. The result will be selected from an average of five trials. Participants can rest between trials for about 2 minutes or as long as they desired to avoid fatigue.
Montreal Cognitive Assessment | Baseline, post-intervention at week 5, 1-month and 3-month after post-intervention
  The MoCA-Thai version will be used to assess cognitive function. All participants will be tested for all domains excepting executive function and visuospatial ability since some participants may unable to complete the written portion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No